CLINICAL TRIAL: NCT06842992
Title: A Multicenter, Randomized, Double-blind, Double-dummy, Placebo and Active-controlled, Dose-exploration Phase II Clinical Trial to Evaluate the Efficacy and Safety of NH102 in the Treatment of Depression
Brief Title: A Phase II Study to Evaluate NH102 for Depression
Acronym: NH102-21
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Nhwa Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NH102-21
Record Dates: First submitted 2025-02-16; First posted 2025-02-24 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Major Depressive Disorder (MDD)
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- NH102 10mg (Experimental)
  Interventions: Drug: NH102
- NH102 20mg (Experimental)
  Interventions: Drug: NH102
- NH102 30mg (Experimental)
  Interventions: Drug: NH102
- Duloxetine Hydrochloride Enteric Capsules (Active Comparator)
  Interventions: Drug: Duloxetine Hydrochloride Enteric-coated Capsule
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NH102 — 5 mg twice daily over 6 weeks, followed by a 1-week tapering period.
  Arms: NH102 10mg
Drug: NH102 — 10 mg twice daily over 6 weeks, followed by a 1-week tapering period.
  Arms: NH102 20mg
Drug: NH102 — 15 mg twice daily over 6 weeks, followed by a 1-week tapering period.
  Arms: NH102 30mg
Drug: Duloxetine Hydrochloride Enteric-coated Capsule — 30 mg twice daily for 6 weeks, followed by a 1-week tapering period.
  Arms: Duloxetine Hydrochloride Enteric Capsules
Drug: Placebo — Matched dosing regimen.Twice daily for 6 weeks, followed by a 1-week tapering period.
  Arms: Placebo

SUMMARY:
This study is a multicenter, randomized, double-blind, double-dummy, parallel-group, dose-finding Phase II clinical trial with placebo and active comparator duloxetine . It is designed to preliminarily assess the efficacy and safety of NH102 in patients with major depressive disorder and to provide the basis for the design of Phase III clinical trials.

DETAILED DESCRIPTION:
This trial consists of three periods: a screening period (up to 2 weeks), a double-blind treatment period (6 weeks), and a tapering-off period/safety follow-up (1 week). The screening period may last up to 14 days and a minimum of 1 day.

Baseline assessments will be conducted prior to randomization to confirm the eligibility of participants. A total of 240 patients with depression will be randomly assigned in a 1:1:1:1:1 ratio to three experimental drug groups (10 mg, 20 mg, and 30 mg), one active control group (duloxetine hydrochloride capsules 60 mg ), or one placebo group. The double-blind treatment period will last for 6 weeks, during which participants will take the assigned medications according to the specified dosing regimen and will be followed up at the end of weeks 1, 2, 4, and 6. After the treatment period, participants will enter a 1-week tapering-off period and will undergo safety follow-up at the end of week 7.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients aged 18-65 years (inclusive).
* Diagnosis of Major Depressive Disorder (MDD) according to DSM-5 criteria ( without psychotic features).
* Hamilton Depression Rating Scale (HAM-D17) total score ≥ 22 at screening and baseline visits, with item 1 (depressed mood) score ≥ 2.
* Clinical Global Impression-Severity (CGI-S) score ≥ 4 at screening and baseline.
* Negative pregnancy test for women of childbearing potential.
* Willingness to use effective contraception during the trial and for 3 months after the last dose.
* Voluntary participation and signed informed consent.

Exclusion Criteria:

* Duration of the current depressive episode in first-episode patients < 3 months.
* Treatment-resistant depression (failure of ≥ 2 adequate antidepressant treatments).
* Other psychiatric disorders (e.g., schizophrenia, bipolar disorder, anxiety disorders).
* History of severe neurological diseases, epilepsy, or significant head trauma.
* Unstable or severe cardiovascular, gastrointestinal, or endocrine diseases.
* History of malignancy within the past 2 years.
* History of increased intraocular pressure or untreated narrow-angle glaucoma.
* Abnormal thyroid function not adequately controlled.
* History of severe drug allergies or hypersensitivity to duloxetine or excipients.
* Suicide attempt within the past year or significant suicide risk.
* Substance abuse within the past year or positive at screening drug test.
* Alcohol abuse (≥ 14 units/week) within the past year.
* Previous treatment with duloxetine without adequate response.
* Normative use of antidepressants within 2 weeks prior to screening.
* Use of CYP2D6 or CYP1A2 potent inhibitors/inducers within 2 weeks prior to screening.
* Participation in another clinical trial within the past 3 months.
* Any condition deemed unsuitable by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2024-12-04 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-09-12 (Actual)

PRIMARY OUTCOMES:
17 items Hamilton Depression Scales (HAM-D17) | 6 Weeks
  Changes from baseline in the 17 items Hamilton Depression Scales (HAM-D17) total score at the end of treatment.
  HAM-D17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression (symptoms such as depressed mood, guilty feelings, suicide, sleep disturbances, anxiety levels, and weight loss). Nine items are scored on a 3 point scale (0=none/absent to 2=most severe) and 8 items are scored on a 5 point scale (0=none/absent to 4=most severe) for a maximum total score of 50. Higher scores indicate a worse outcome.

SECONDARY OUTCOMES:
17 items Hamilton Depression Scales (HAM-D17) | Week 2 and 4
  Changes from baseline in the 17 items Hamilton Depression Scales (HAM-D17) total score at Week 2 and 4.
  HAM-D17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression (symptoms such as depressed mood, guilty feelings, suicide, sleep disturbances, anxiety levels, and weight loss). Nine items are scored on a 3 point scale (0=none/absent to 2=most severe) and 8 items are scored on a 5 point scale (0=none/absent to 4=most severe) for a maximum total score of 50. Higher scores indicate a worse outcome.
Montgomery- Åsberg Depression Rating Scale(MADRS) | 6 Weeks
  Changes from baseline in the 10-items Montgomery- Åsberg Depression Scales (MADRS) total score at Week 2, Week 4 and the end of treatment.
  MADRS is a standardized, clinician-administered rating scale that assesses 10 items characteristically associated with major depression. Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms).
Clinical Global Impression-Improvement (CGI-I) | 6 Weeks
  Changes from baseline in the CGI-I score at the end of treatment.
  The Clinical Global Impression-Improvement (CGI-I) scale is a clinician-rated instrument designed to assess the overall improvement or worsening of a patient's condition relative to a baseline state. The following one query is rated on a seven-point scale: "Compared to the patient's condition at admission to the project, this patient's condition is: 1=very much improved since the initiation of treatment; 2=much improved; 3=minimally improved; 4=no change from baseline (the initiation of treatment); 5=minimally worse; 6= much worse; 7=very much worse since the initiation of treatment."
Clinical Global Impression-Severity (CGI-S) | 6 Weeks
  Changes from baseline in the Clinical Global Impression-Severity (CGI-S) score at the end of treatment.
  The CGI-S asks the clinician one question: "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?" which is rated on the following seven-point scale: 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients.
Hamilton Anxiety Rating Scale (HAM-A) | 6 Weeks
  Changes from baseline in the HAM-A total score at the end of treatment.
  The Hamilton Anxiety Rating Scale (HAM-A) is a clinician-administered assessment tool to measure the severity of anxiety symptoms. It consists of 14 items, each evaluating a specific symptom of anxiety, such as anxious mood, tension, fears, and somatic complaints. Each item is scored on a scale from 0 (None) to 4 ( Very severe. grossly disabling ), with the total score ranging from a minimum of 0 to a maximum of 56. Higher scores indicate greater severity of anxiety symptoms, reflecting a worse clinical outcome.
Dimensional Anhedonia Rating Scale (DARS) | 6 Weeks
  Change from baseline in Dimensional Anhedonia Rating Scale (DARS) total score at the end of treatment.
  The DARS is a self-report scale that measures anhedonia across the following 4 domains: hobbies/past-times, food/drinks, social activities, and sensory experiences. Within each domain, participants are required to provide at least two of their own examples of what they find rewarding. Subsequently, participants answer a set of standardized questions about desire, motivation, effort and consummatory pleasure for the examples provided. Responses were based on a 5-point Likert scale (Not at all=0; Slightly=1; Moderately=2; Mostly=3; Very Much=4), with the total score ranging from a minimum of 0 to a maximum of 68. A higher score reflects a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided